CLINICAL TRIAL: NCT00742573
Title: Improving the Effectiveness of Treatment for Depression in Hispanics
Brief Title: Incorporating Patient Treatment Choice to Improve Treatment Retention in Depressed Hispanics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mark Olfson, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #5692; R01MH076051 (NIH); DSIR 83-ATSO
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Mood Disorders; Hispanic
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders | interventions — Citalopram; Escitalopram; Paroxetine; Sertraline; Venlafaxine Hydrochloride; Bupropion; Duloxetine Hydrochloride; Nortriptyline; Mirtazapine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Texas Medication Algorithm (Active Comparator): Participants will receive medication treatment according to the Texas Medication Algorithm (TMA) for depression
  Interventions: Drug: Antidepressants through Texas Medication Algorithm (TMA)
- 2 Patient Choice (Experimental): Participants will be offered brief interpersonal psychotherapy (IPT-B) alone or combined with the TMA for depression
  Interventions: Drug: Antidepressants through Texas Medication Algorithm (TMA); Behavioral: Brief Interpersonal Psychotherapy (IPT-B)

INTERVENTIONS:
Drug: Antidepressants through Texas Medication Algorithm (TMA) — Treatment with medication will follow the TMA for depression. Antidepressant medications may include any of the following: citalopram, escitalopram, paroxetine, sertraline, venlafaxine XR, bupropion SR, duloxetine, nortriptyline, and mirtazapine.
  Other Names: Celexa; Lexapro; Paxil; Zoloft; Effexor XR; Wellbutrin; Cymbalta; Pamelor; Remeron
Behavioral: Brief Interpersonal Psychotherapy (IPT-B) — IPT-B consists of twelve 50-minute sessions, divided into three phases, focusing on an interpersonal problem or problems.
  Arms: 2 Patient Choice

SUMMARY:
This study will determine whether combination treatment driven by patient choice is better than standardized medication treatment at retaining and improving Hispanic patients with major depressive disorder.

DETAILED DESCRIPTION:
Retention of Hispanics in the treatment of major depressive disorder (MDD) continues to be a major public health problem. Hispanics drop out from treatment two to three times more frequently than non-Hispanic whites, despite the scarcity of treatment alternatives for Hispanics and their low rates of re-entry into the mental health care system. Consistent with the goals of Healthy People 2010 and the President's New Freedom Commission on Mental Health, the goal of this study is to test the efficacy in a research setting of a novel intervention to improve retention and response. This efficacy assessment would serve as a reference point for the development of future effectiveness trials in community settings.

Our intervention is founded on growing evidence that when depressed Hispanics seek help for mental health problems, they prefer to receive psychotherapy or combined treatment in the form of weekly in-person clinic visits. However, socioeconomic barriers, such as low-paying jobs with irregular hours, lack of child care, and limited time availability, often reduce treatment retention and result in dropout rates up to three times those of non-Hispanic whites. Based on emerging literature and on promising pilot data, we propose to study the efficacy for depressed Hispanics of an intervention that would allow for patient choice between the following options: 1) Medication alone, following the Texas Medication Algorithm for Depression (TMA); 2) Brief Interpersonal Psychotherapy (IPT-B) alone, with optional telephone sessions; or 3) Combined medication plus IPT-B. This intervention would allow switching of treatment modality (e.g., from IPT-B alone to combined treatment) at any point during the study period. We hypothesize that by permitting patient choice among evidence-based treatments, flexibility in the sequential use of treatments, and novel treatment delivery systems, this intervention will substantially increase retention of Hispanics in MDD treatment. Furthermore, we will examine mediators and moderators of retention, including stigma and insurance coverage.

We propose to test this intervention in depressed Hispanics seeking outpatient psychiatric treatment using a randomized trial with TMA as the control group. Both groups will have access to medication using the TMA but only one group will be offered IPT_B. . We will test the association between treatment, retention, and response over the course of acute MDD care (12 weeks), and will also obtain preliminary outcome data after 9 more months of treatment (i.e., for a total of 12 months). Our pilot data enable us to estimate the sample size for the acute phase, while the additional follow-up period allows us to examine the effect of choice over the longer-term course of MDD care.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic males and females
* DSM-IV criteria for non-psychotic major depressive disorder (MDD) of at least moderate severity (HAM-D-17> 18)
* 18- 79
* Patients with stable dosage of Benzodiazepines to treat anxiety disorders

Exclusion Criteria:

* At risk of attempting suicide
* Unstable medical illness
* History of bipolar disorder, schizophrenia, or other psychotic disorder
* Pregnant or lactating
* Alcohol or substance use disorder that requires acute detoxification

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2008-08; Primary Completion 2014-01-10 (Actual); Study Completion 2014-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Blanco, MD, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant available to other researchers at this time.

REFERENCES:
- [Derived] Blanco C, Markowitz JC, Hellerstein DJ, Nezu AM, Wall M, Olfson M, Chen Y, Levenson J, Onishi M, Varona C, Okuda M, Hershman DL. A randomized trial of interpersonal psychotherapy, problem solving therapy, and supportive therapy for major depressive disorder in women with breast cancer. Breast Cancer Res Treat. 2019 Jan;173(2):353-364. doi: 10.1007/s10549-018-4994-5. Epub 2018 Oct 20. PMID 30343455

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 Texas Medication Algorithm | 2 Patient Choice
Started | 83 | 87
Week 12 | 46 | 51
Week 24 | 39 | 37
Week 52 | 26 | 25
Completed | 26 | 25
Not Completed | 57 | 62

BASELINE CHARACTERISTICS:
Population: Adult Hispanics with MDD
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Texas Medication Algorithm | 2 Patient Choice | Total
Number analyzed (Participants) | 83 | 87 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 79 | 85 | 164
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (12.5) | 40.8 (11.2) | 39.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 35 | 38 | 73
Region of Enrollment [Number; unit: participants]
  United States | 83 | 87 | 170

OUTCOME MEASURES:

1. Primary Outcome: Mean Time of Retention
Description: Average number of weeks of retention of Hispanics in the treatment of MDD
Time Frame: 52 weeks
Population: Adult Hispanics with MDD
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | 1 Texas Medication Algorithm | 2 Patient Choice
Number analyzed (Participants) | 83 | 87
weeks | 27.08 (22.4) | 25.84 (20.54)

2. Primary Outcome: Hamilton Depression Scale (HAMD-17)
Description: Hamilton Depression Scale (HAMD-17): Scoring is based on the 17-item scale of 0-4, the higher the worse.
  0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression, over 24 severe depression
  Minimum is 0 and the maximum score being 52
Time Frame: Baseline
Population: Adult Hispanics with MDD and Non-missing HAMD Total Score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1 Texas Medication Algorithm | 2 Patient Choice
Number analyzed (Participants) | 37 | 38
score on a scale | 23.89 (3.96) | 22.42 (3.64)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | 1 Texas Medication Algorithm | 2 Patient Choice
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/87
Other Adverse Events (participants affected / at risk) | 0/83 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes